CLINICAL TRIAL: NCT00815477
Title: I-START: Internet-based Strategic Transdisciplinay Approach to Risk Reduction And Treatment
Brief Title: Internet-Based Strategic Transdisciplinary Approach To Risk Reduction And Treatment
Acronym: I-START
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Stroke Network (Other)
Responsible Party: Principal Investigator, Robert Nolan, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06-0422-BE; Candian Stroke Network
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Waitlist control with generic Information about lifestyle and hypertension
  Interventions: Behavioral: Generic Information
- 2 (Experimental): Web-based intervention of lifestyle counseling messages based on the transtheoretical model of readiness for change.
  Interventions: Behavioral: Web-based lifestyle counseling messages

INTERVENTIONS:
Behavioral: Web-based lifestyle counseling messages — 10 email messages based on readiness-to-change over a 4 month period
  Arms: 2
Behavioral: Generic Information — Waitlist control plus educational material on lifestyle behavior and hyptertension
  Arms: 1

SUMMARY:
I-START is a randomized controlled trial that will evaluate the efficacy of an internet-based program of behavioural counseling for adaptive lifestyle change to subjects diagnosed with hypertension. I-START will be evaluated using objective outcome indices: systolic and diastolic blood pressure, pulse pressure, and markers of vagal-heart rate (HR) modulation and baroreflex sensitivity. The Heart and Stroke Foundation of Canada "Blood Pressure Action Plan(TM)" (BPAP) will be adminisered over a 4-month period, and evaluated in a 2 (Intervention vs. Wait list Control) X 2 (Baseline vs. Post-Intervention) factorial design, blocking for 3 recruitment sites (Toronto, London, the Grey Bruce region of Ontario, Canada), and stratified for sex and age group (45-59, 60-74 years).

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 OR Stage 2 hypertension
* 46 -74 years of age
* able to read & write English or French
* living in private residence

Exclusion Criteria:

* Cardiovascular disease
* Major psychiatric disorder (e.g. psychosis)
* Dependence on Alcohol or Drugs with in past year
* Diabetes >= 5 years

Ages: 46 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Lab Assessment of systolic and diastolic blood pressure as well as pulse pressure | 4 months

SECONDARY OUTCOMES:
Lifestyle Behavior: exercise and diet assessed by questionnaire | 4 months
laboratory assessment of estimated vagal-heart rate modulation and baroreflex sensitivity | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Nolan, Ph.D., Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - University of Western Ontario, London, Ontario
  - Grey Bruce Public Health Unit, Owen Sound, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Result] Durrani S, Irvine J, Nolan RP. Psychosocial determinants of health behaviour change in an e-counseling intervention for hypertension. Int J Hypertens. 2012;2012:191789. doi: 10.1155/2012/191789. Epub 2011 Dec 20. PMID 22229083
- [Derived] Nolan RP, Liu S, Shoemaker JK, Hachinski V, Lynn H, Mikulis DJ, Wennberg RA, Moy Lum-Kwong M, Zbib A. Therapeutic benefit of internet-based lifestyle counselling for hypertension. Can J Cardiol. 2012 May;28(3):390-6. doi: 10.1016/j.cjca.2012.02.012. Epub 2012 Apr 11. PMID 22498181